CLINICAL TRIAL: NCT03947580
Title: Clinical Trial Evaluating the Effectiveness and Safety of Dvectis Single and Dvectis Double Pads in Comparison to "no Pad Use" in Patients With Chronic Lumbar Spine Pain
Brief Title: Clinical Trial of Dvectis Pads in Comparison to no Pad Use in Patients With Chronic Lumbar Spine Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DD-Hippero s.r.o. (Industry)
Collaborators: PharmTest s.r.o. (Industry); Prague Clinical Services s.r.o. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DVE-17
Record Dates: First submitted 2019-04-11; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-04

CONDITIONS: Back Pain; Back Disorder; Disease Lumbar Spine
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Use of the Dvectis Single pad (Experimental): The Dvectis Single Dynamic-directional pad is a basic model of the Dvectis product range that provides full functionality based on the dynamic-directional seating principle. The Dvectis Single pad is designed to steer muscle tension during sitting in deep-seated muscles. The Dvectis Single pad is intended to eliminate chronic lumbar spine pain by strengthening the stabilizing muscles.
  Interventions: Other: Use of the Dvectis Single pad; Other: Use of no pad
- Use of the Dvectis Double pad (Experimental): The Dvectis Double Dynamic-directional pad is based on the Dvectis Single model, but in addition to its dual-chamber design, it provides seating with a more balanced load and a higher dynamic-directional effect. The Dvectis Double pad is designed to create and route muscle tension during sitting in deep-seated muscles. The Dvectis Double is also suitable for soft substrates (sofa, soft chair, etc.). The Dvectis Double Pad is intended to remove chronic lumbar spine pain by strengthening the stabilizing muscles.
  Interventions: Other: Use of the Dvectis Double pad; Other: Use of no pad
- Use of no pad (No Intervention): Description is not needed

INTERVENTIONS:
Other: Use of the Dvectis Single pad — Change in pain intensity - range of VAS (mm) between Visit 1 and Visit 2 Dvectis Single pads compared to "without using a pad".
  Arms: Use of the Dvectis Single pad
Other: Use of the Dvectis Double pad — Change in pain intensity - range of VAS (mm) between Visit 1 and Visit 2 Dvectis Double pad compared to "without using a pad",
  * Categorisation of adverse events,
  * Categorisation of deficiencies of a medical device in patients enrolled in treatment groups using Dvectis Single and Dvectis Double pad,
  * Number of patients with adverse events,
  * Number of patients with deficiencies of medical device enrolled in treatment groups using Dvectis Single and Dvectis Double
  Arms: Use of the Dvectis Double pad
Other: Use of no pad — Description is not needed
  Arms: Use of the Dvectis Double pad; Use of the Dvectis Single pad

SUMMARY:
1. Introduction

1.1 Description of the Trial

The trial was a monocentric, open, randomized, 3-arm clinical trial that took place at the Department of Orthopaedics of the Karviná Miners' Hospital (Karvinská hornická nemocnice a.s.). The involvement of a maximum total number of 198 patients with chronic lumbar spine pain was planned; the patients were randomly and evenly assigned to one of the 3 treatment groups:

1. Use of the Dvectis Single pad;
2. Use of the Dvectis Double pad;
3. Use of no pad. One sequential interim analysis was planned in the middle of the clinical trial and after this interim analysis, the trial was stopped early due to proven efficacy.

The expected period of participation of each patient in the clinical trial was 6 weeks (± 5 days). For an overview of the individual study visits and procedures, study population and other detailed information, see the study protocol.

According to the plan, the assessment subject was asked during Visit 1 and Visit 2 about the most intensive pain felt in the last 48 hours (PI). The pain was recorded by the subject in the visual analogue scale (VAS) in CRF under supervision of the investigator. Then the assessment subject recorded the intensity of their pain independently in the Patient Journal daily.

1.2 Primary Objective, Quantity and Hypothesis

The primary objective of the clinical trial was to assess the efficacy of using the Dvectis Single pad in comparison to "use of no pad" in patients suffering from chronic lumbar spine pain.

PI was the primary quantity. The primary hypothesis was the superiority of Dvectis Single based on a check, assessed based on the difference in PI (PID) between week 2 and week 6 (PID6).

DETAILED DESCRIPTION:
1. Analysed Populations and Number of Subjects

Prior to the statistical analysis, 4 populations were defined in line with the study protocol:

1. Population including all randomised subjects (ARS);
2. Population of all patient with intention to treat (ITT);
3. Population of patients without serious deviation from the clinical trial plan
4. Safety population.

Each analysed population was based on a list of its members. Although the treatment group could have generally been different for each patient in a different population (see the study protocol and statistical analysis plan), such a case did not occur (as all the patients were de facto placed in the group to which they were randomized). Therefore the real treatment group is the same as the randomization treatment group for all patients. This fact is not discussed further in the document.

1.1 The ARS population

Included all patients who were involved in the clinical trial and randomized. The ARS population was used for summaries of demographic quantities and other quantities established during Visit 1 in order to describe the study population.

1.2 ITT Population

In this case, this population was identical to the ARS population. According to the plan, ITT was not supposed to include those ARS patients for whom no PI data were available and those patients who entered the study repeatedly. However, such circumstances were not detected. The ITT population represented the primary analysed population for the assessment of efficacy.

1.3 PPS Population

According to the statistical plan, PPS was to include all ITT patients except for patients with a serious deviation from the clinical trial plan; a serious deviation includes:

* Failure to meet one or multiple participation criteria;
* Error in treatment allocation;
* Documented use of unauthorized concomitant medication or treatment;
* Missing PI0 value;
* More than 25% missing PI values.
* Serious treatment regimen violation or another serious deviation from the clinical trial plan.

The monitoring reports and discrepancy report implied:

* No study subject that has not met a participation criterion has been registered;
* No study subject with incorrectly allocated treatment has been identified;
* No use of unauthorized concomitant treatment has been documented;
* There was no PI0 value missing;
* Patients 45, 53 and 94 ended the study early; the number of PI values missing is over 25% (83%).
* The following patients violated the treatment regimen in terms of non-observance of the minimum time of sitting on the pad (21, 23, 35, 42, 55, 57, 60, 72, 75, 76, 84, 86, 88).

Thus there was a serious deviation from the protocol in 16 study subject, i.e. 15.7%.

The PPS population represented the secondary analyzed population for the assessment of efficacy. Its task was to demonstrate the robustness of the main clinical trial results. For this reason, comparisons of the tested group efficacy to the control group were used (in addition to ITT) in final analyses using PI in order to achieve confirmation of the main clinical trial conclusions.

1.4 Safety Population

According to the plan, the safety population should have constituted of subjects from ARS, except for those with whom all contact was lost immediately after Visit 1 and those who were placed (in reality) in one of the tested groups but were not given a pad.A pad was given to all patients in the tested groups. All contact was lost with patients 53 and 94 and they were eliminated from the safety population. Patients in the safety population were analyzed based on the treatment groups they were really placed in, regardless of what group they had been randomized to.

1.6. Overview of Analysed Populations and Patient History (Numbers of subjects in treatment groups and analysed populations)

Dvectis Dvectis No treatment Total Single Double

ARS population 35 34 33 102 ITT population 35 34 33 102 PPS population 29 25 32 86 Safety population 35 33 32 100

2 Missing Data

In the ARS population analyses, the missing data were be treated as missing according to the plan, i.e. stated in summaries as total numbers of missing data; however, they were excluded from the calculations of other statistics. In reality, only the time of sitting on the pad is of significance. In all analyses of the PI quantities, the method of imputation of the last observed value (Last Observation Carried Forward - LOCF) was used, in accordance with the plan. The plans for a situation when the PI1 would be missing were not used since the situation did not occur. The use of LOCF generally also leads to a bias but with regard to the observed decrease in the PI values during the patient's participation in the study in the tested groups, compared to the reference group, such an approach is obviously conservative. For evaluation of the Oswestry questionnaire, the use of LOCF was planned primarily at the level of individual questions as well as the use of the scoring manual procedure accounting for missing values, if any. This procedure was beyond the data administration and statistical analysis activities since the questionnaire was evaluated by the investigator, entering only the total score in the patient record sheets. If the total score was missing, it was processed similarly to the processing of missing values in the ARS population analysis (i.e. solely elimination from the analysis).

3 Sequential and Final Analysis

The first sequential analysis was performed according to the interim analysis plan and resulted in early study stopping due to efficacy. A report of the first sequential analysis results is included in a separate document. Then the final analysis was performed, which is presented in this report.

4 Characteristic of Study Subject and Treatment Regimen Compliance

For the description of the study population within the sequential interim analysis, summaries of demographic quantities were calculated and presented, as established before the start of the treatment in the scope determined by the statistical analysis plan. The summaries were presented for the respective treatment groups (for all 3 treatment groups). The significance of the differences in these characteristics was not tested.

The treatment regimen compliance was evaluated by a calculation of aggregate statistics for the average time of the device use in the course of participation in the study.

For the analyzed quantities, summary statistics were calculated in the respective treatment groups and as a total. The analyzed ARS population was used.

ELIGIBILITY:
* inclusion criteria:

  1. Age 18-65 years.
  2. The Condition of chronic musculoskeletal pain in the lumbar spine (degenerative diseases of the spine) for at least the last 3 months without a major change in the intensity of pain.
  3. VAS ≥ 40 mm of lumbar spine pain felt in the last 48 hours.
* exclusion criteria:

  1. Chronic pain caused by diseases other than degenerative diseases of the spine.
  2. Any condition/disease or medicine found in the medical history of the screening, which in the investigator's opinion could affect the assessment of the intensity of pain.
  3. Physiotherapeutic rehabilitation in the spine planned at the time of participation in the clinical test.
  4. Pregnant or breastfeeding woman.
  5. Simultaneous participation in another clinical investigation or study.
  6. Inability to understand patient Information and unwillingness to cooperate in compliance with the clinical investigation instructions.
  7. Unsigned Informed consent.
* Criteria for early termination of participation:

  1. The subject's wish to end participation.
  2. The Occurrence of non-inclusion criteria during the clinical investigation.
  3. Occurrence of a serious adverse event or other circumstance where further persistence in the clinical investigation would endanger the subject's health.
  4. Impossibility to comply with the clinical investigation plan, e.g. Insufficient compliance with the guidelines by the subject or for organisational reasons.
  5. Deterioration of the subject's health status, which will require unauthorised treatment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Change of pain intensity of using the Dvectis Single pad in comparison to "use of no pad" in patients at Visit 1 and Visit 2 | 6 weeks between visits
  Pain intensity was measured on a 100 mm Visual Analogue Scale (VAS). VAS is a graphic record where the patient indicates the intensity of pain on a 100 mm long line, where 0 mm means no pain and 100 mm means unbearable pain. The degree of pain intensity is the distance from the left end of the line to the patient indicated by the value in millimeters. The participating subject was asked for experiencing the greatest pain in the last 48 hours during the Visit 1 and Visit 2. The pain was recorded by the subject under supervision of the investigator at Visit 1 and Visit 2. Change of VAS values in mm (0-100mm) between Visit 1 and 2 was evaluated for all subjects. Finaly the overall changes of pain intensity of patients using the Dvectis Single pad in comparison to "use of no pad" were evaluated by statistician.

SECONDARY OUTCOMES:
Change of pain intensity of using the Dvectis Double pad in comparison to "use of no pad" in patients at Visit 1 and Visit 2 | 6 weeks between visits
  Pain intensity was measured on a 100 mm Visual Analogue Scale (VAS). VAS is a graphic record where the patient indicates the intensity of pain on a 100 mm long line, where 0 mm means no pain and 100 mm means unbearable pain. The degree of pain intensity is the distance from the left end of the line to the patient indicated by the value in millimeters. The participating subject was asked for experiencing the greatest pain in the last 48 hours during the Visit 1 and Visit 2. The pain was recorded by the subject under supervision of the investigator at Visit 1 and Visit 2. Change of VAS values in mm (0-100mm) between Visit 1 and 2 was evaluated for all subjects. Finaly the overall changes of pain intensity of patients using the Dvectis Double pad in comparison to "use of no pad" were evaluated by statistician.

OTHER OUTCOMES:
Number and categorization of adverse events of each patient | 6 weeks
  Number and categorization of adverse events are evaluated by Principal investigator and recorded in Case Report Form (CRF) for each patient. No scale is used. Categorization is - serious or not serious adverse event. Categorization is done at Visit 1 and Visit 2.
Number and categorization of deficiencies of the medical device in patients enrolled in treatment groups using Dvectis Single or Dvectis Double pad | 6 weeks
  Number and categorization of deficiencies of the medical device are evaluated by Principal investigator and recorded in Case Report Form (CRF) for each patient. No scale is used. Categorization is - mechanical damage, manufacturing defect, other (descriptive). Categorization is done at Visit 1 and Visit 2.
Number of patients with adverse events | 6 weeks (one patient)
  Number of patients with adverse events. The number is summarized and evaluated by statistician at the end of experimental phase of the study.
Number of patients with deficiencies of the medical device | 6 weeks (one patient)
  Number of patients with deficiencies of the medical device. The number is summarized and evaluated by statistician at the end of experimental phase of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Marietta Tesarova, MUDr., Study Chair — prague clinical services
Locations (1):
- Prague Clinical Services, Prague, Praha 4, Czechia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT03947580/Prot_SAP_000.pdf